CLINICAL TRIAL: NCT03753581
Title: Effectiveness of Microcurrents Therapy in Pressure Ulcers in Elderly People: Controlled and Randomized Triple Blind Clinical Trial
Brief Title: Effectiveness of Microcurrents Therapy in Pressure Ulcers in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Residencia Geriátrica San Diego, S.L. (Unknown); Residencia de Mayores Río Tajo ARTEVIDA. Centro Serviger Talavera (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EUEYF
Record Dates: First submitted 2018-10-04; First posted 2018-11-27 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2018-11

CONDITIONS: Electric Stimulation Therapy
Keywords: Electric Stimulation Therapy; Pressure Ulcer; Aged
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Masking of the researchers: the assignment of participants to the groups will be carried out by a researcher who will not apply the interventions and will not collect the outcome variables. The interventions will be carried out by researchers different from those who will perform the evaluations of the outcome variables.
  Masking of the participants: it will be done using the same electrodes and microcurrent devices in both groups. In the placebo stimulation, the device will emit a luminous signal of operation as well as the devices of the intervention group, however, it will be manipulated and tested with an oscilloscope to ensure that it does not emit microcurrents. The participants of both groups will not perceive any sensation of current, since the electrical stimulation with microcurrents is below the sensitive threshold.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care protocol plus microcurrents (Experimental): * Standardized protocol of nursing care: postural treatment plus standardized cure.
  * Intervention with microcurrents: application of 2 electrodes (Mc Patch, Newmark USA) around the ulcer.
  Interventions: Device: Care protocol plus microcurrents
- Care protocol plus placebo microcurrents (Placebo Comparator): * Standardized protocol of nursing care: postural treatment plus standardized cure.
  * Placebo microcurrents: application of 2 electrodes (Mc Patch, Newmark USA) around the ulcer previously handled that do not emit current.
  Interventions: Device: Care protocol plus placebo microcurrents

INTERVENTIONS:
Device: Care protocol plus microcurrents — CARE NURSING PROTOCOL: postural treatment every 4 hours more standardized cure according to the guide of recommendations based on evidence in prevention and treatment of pressure ulcers in adults of Osakidetza health service.
  MICROCURRENTS: the electrodes will be placed on the edge of the dressing on the sides of the ulcer's longer length during 12 hours a day until the ulcer is completely healed or for a maximum of 25 days.
  Characteristics of microcurrents: pulsed monophasic rectangular wave with a pulse of 1.5 s and pause of 300 ms, voltage 21 mV and intensity 42μA with a current density of 4.2 μA.
  Arms: Care protocol plus microcurrents
Device: Care protocol plus placebo microcurrents — The same nursing care protocol described for the experimental group will be applied more 12 hours per day of 2 electrodes of microcurrents around the ulcer, which will be previously manipulated and tested with an oscilloscope so that they do not emit electrical currents
  Arms: Care protocol plus placebo microcurrents

SUMMARY:
The purpose of this study is to investigate the effect on the healing of pressure ulcers in elderly people using a care protocol plus the application of microcurrent patches during 12 hours per day compared to the effect of the same protocol plus placebo electric stimulation.

DETAILED DESCRIPTION:
The design of this study is a multicentric, parallel, randomised, triple blind clinical trial with placebo control.

The size of the sample will be 30 participants older than 60 years old who are institutionalized in some nursing homes in Spain.They will be randomized in two groups: control or experimental.

The variables of the study will be collected at three time points: before the intervention, 14 days after the start of the intervention and at the end of the intervention.

The statistical analysis will be an intention-to-treat analysis. For the main outcomes variables a two-factor ANOVA will-be performed (intervention-time) with a post-hoc analysis with Bonferroni correction

ELIGIBILITY:
Inclusion Criteria:

* Adults over 60 institutionalized in nursing homes.
* Participants presenting pressure ulcers in phase II, III and IV according to the North American National Pressure Ulcer Advisory Panel System and the European Pressure Ulcer Advisory Panel System.
* Time of evolution of the pressure ulcer greater than 1 month and less than 24 months.
* Ulcer size greater than 1 cm2.
* Less than 14 points on the Braden scale.

Exclusion Criteria:

* Presence of a pacemaker or any implanted electrical device.
* Metal implants in the pressure ulcer area.
* Pressure ulcer in occipital area.
* Cancer.
* Osteomyelitis.
* 3 or more abnormal blood values at the beginning of the study that indicate a limited healing potential (anemia, iron deficiency, protein deficiency, dehydration, uncontrolled diabetes or hypothyroidism)
* Allergies to the usual cures protocol established.
* Systemic infection
* Recent history (minimum of 30 days) of treatment with growth factors or vacuum-assisted treatment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Ulcer healing 1 day before the intervention start | 1 day before the start of the intervention
  It will be evaluated with the Pressure Ulcer Scale for Healing (PUSH). It was developed by the National Pressure Ulcer Advisory Panel (NPUAP) to monitor the change in the status of pressure ulcers over time.
  The ulcer is categorized according to the surface area, exudate and type of wound tissue. A partial score is recorded for each of these ulcer characteristics:
  * Surface area (in cm2): 10 points (0 points=0 cm2; 10 points= >24 cm2)
  * Exudate amount: 3 points (0 points= none; 3 points=heavy).
  * Tissue type: 4 points (0 points= closed; 4 points= necrotic tissue).
  To obtain the total score, the sub-scores are added. The minimum score is 0, which means that the ulcer is healed and the maximum score is 17, which means that the ulcer surface is greater than 24 cm2, that there is a heavy exudate and necrotic tissue.
  A comparison of total scores measured over time provides an indication of the improvement or deterioration in pressure ulcer healing.
Ulcer healing at 14 days | At 14 days after the start of the intervention
  It will be evaluated with the Pressure Ulcer Scale for Healing (PUSH). It was developed by the National Pressure Ulcer Advisory Panel (NPUAP) to monitor the change in the status of pressure ulcers over time.
  The ulcer is categorized according to the surface area, exudate and type of wound tissue. A partial score is recorded for each of these ulcer characteristics:
  * Surface area (in cm2): 10 points (0 points=0 cm2; 10 points= >24 cm2)
  * Exudate amount: 3 points (0 points= none; 3 points=heavy).
  * Tissue type: 4 points (0 points= closed; 4 points= necrotic tissue).
  To obtain the total score, the sub-scores are added. The minimum score is 0, which means that the ulcer is healed and the maximum score is 17, which means that the ulcer surface is greater than 24 cm2, that there is a heavy exudate and necrotic tissue.
  A comparison of total scores measured over time provides an indication of the improvement or deterioration in pressure ulcer healing.
Ulcer healing at 26 days | At 26 days after the start of the intervention
  It will be evaluated with the Pressure Ulcer Scale for Healing (PUSH). It was developed by the National Pressure Ulcer Advisory Panel (NPUAP) to monitor the change in the status of pressure ulcers over time.
  The ulcer is categorized according to the surface area, exudate and type of wound tissue. A partial score is recorded for each of these ulcer characteristics:
  * Surface area (in cm2): 10 points (0 points=0 cm2; 10 points= >24 cm2)
  * Exudate amount: 3 points (0 points= none; 3 points=heavy).
  * Tissue type: 4 points (0 points= closed; 4 points= necrotic tissue).
  To obtain the total score, the sub-scores are added. The minimum score is 0, which means that the ulcer is healed and the maximum score is 17, which means that the ulcer surface is greater than 24 cm2, that there is a heavy exudate and necrotic tissue.
  A comparison of total scores measured over time provides an indication of the improvement or deterioration in pressure ulcer healing.

SECONDARY OUTCOMES:
Stage of pressure ulcer 1 day before the intervention start | 1 day before the start of the intervention
  According to the North American National Pressure Ulcer Advisory Panel System and the European Pressure Ulcer Advisory Panel System
Stage of pressure ulcer at 14 days | At 14 days after the start of the intervention
  According to the North American National Pressure Ulcer Advisory Panel System and the European Pressure Ulcer Advisory Panel System
Stage of pressure ulcer at 26 days | At 26 days after the start of the intervention
  According to the North American National Pressure Ulcer Advisory Panel System and the European Pressure Ulcer Advisory Panel System
Ulcer depth 1 day before the intervention start | 1 day before the start of the intervention
  It will be registered in mm with a Swab, specimen collection. Deltalab, SL
Ulcer depth at 14 days | At 14 days after the start of the intervention
  It will be registered in mm with a Swab, specimen collection. Deltalab, SL
Ulcer depth at 26 days | At 26 days after the start of the intervention
  It will be registered in mm with a Swab, specimen collection. Deltalab, SL
Ulcer área 1 day before the intervention start | 1 day before the start of the intervention
  It will be registered in cm2 with the application for pressure ulcer management Mobile Wound Analyzer (MOWA) for IOS Version 1.7.2011. Developer: Bello Ciro (Italy)
Ulcer área at 14 days | At 14 days after the start of the intervention
  It will be registered in cm2 with the application for pressure ulcer management Mobile Wound Analyzer (MOWA) for IOS Version 1.7.2011. Developer: Bello Ciro (Italy)
Ulcer área at 26 days | At 26 days after the start of the intervention
  It will be registered in cm2 with the application for pressure ulcer management Mobile Wound Analyzer (MOWA) for IOS Version 1.7.2011. Developer: Bello Ciro (Italy)
Cutaneous blood flow in the area surrounding the pressure ulcer 1 day before the intervention start | 1 day before the start of the intervention
  It will be recorded in the greater side of the ulcer by cutaneous doppler laser flowmetry with a scale of 0-1000 units (model DRT4, Moor instruments, Devon, UK)
Cutaneous blood flow in the area surrounding the pressure ulcer at 14 days | At 14 days after the start of the intervention
  It will be recorded in the greater side of the ulcer by cutaneous doppler laser flowmetry with a scale of 0-1000 units (model DRT4, Moor instruments, Devon, UK)
Cutaneous blood flow in the area surrounding the pressure ulcer at 26 days | At 26 days after the start of the intervention
  It will be recorded in the greater side of the ulcer by cutaneous doppler laser flowmetry with a scale of 0-1000 units (model DRT4, Moor instruments, Devon, UK)
Pain caused by pressure ulcer 1 day before the intervention start: numerical scale | 1 day before the start of the intervention
  It will be assessed with the numerical scale of the pain that includes the values from 0 (absence of pain) to 10 (maximum pain)
Pain caused by pressure ulcer at 14 days: numerical scale | At 14 days after the start of the intervention
  It will be assessed with the numerical scale of the pain that includes the values from 0 (absence of pain) to 10 (maximum pain)
Pain caused by pressure ulcer at 26 days: numerical scale | At 26 days after the start of the intervention
  It will be assessed with the numerical scale of the pain that includes the values from 0 (absence of pain) to 10 (maximum pain)
Administration of analgesic drugs 1 day before the intervention start | 1 day before the start of the intervention
  The type of analgesic will be registered according to WHO therapeutic steps
Administration of analgesic drugs at 14 days | At 14 days after the start of the intervention
  The type of analgesic will be registered according to WHO therapeutic steps
Administration of analgesic drugs at 26 days | At 26 days after the start of the intervention
  The type of analgesic will be registered according to WHO therapeutic steps
Exudate culture of the ulcer 1 day before the intervention start | 1 day before the start of the intervention
  The presence of infection in the ulcer will be evaluated with a exudate culture
Exudate culture of the ulcer at 14 days | At 14 days after the start of the intervention
  The presence of infection in the ulcer will be evaluated with a exudate culture
Exudate culture of the ulcer at 26 days | At 26 days after the start of the intervention
  The presence of infection in the ulcer will be evaluated with a exudate culture
Administration of systemic antibiotics 1 day before the intervention start | 1 day before the start of the intervention
  The administration of antibiotics will be recorded
Administration of systemic antibiotics at 14 days | At 14 days after the start of the intervention
  The administration of antibiotics will be recorded
Administration of systemic antibiotics at 26 days | At 26 days after the start of the intervention
  The administration of antibiotics will be recorded
Blood pressure 1 day before the intervention start | 1 day before the start of the intervention
  The systolic and diastolic blood pressure will be recorded in mm/Hg with a tensiometer. It will be taken at rest, making 2 measurements separated by a 1-2 minute interval
Blood pressure at 14 days | At 14 days after the start of the intervention
  The systolic and diastolic blood pressure will be recorded in mm/Hg with a tensiometer. It will be taken at rest, making 2 measurements separated by a 1-2 minute interval
Blood pressure at 26 days | At 26 days after the start of the intervention
  The systolic and diastolic blood pressure will be recorded in mm/Hg with a tensiometer. It will be taken at rest, making 2 measurements separated by a 1-2 minute interval
Capillary blood glucose 1 day before the intervention start | 1 day before the start of the intervention
  It will be recorded in mg/dl with a glucometer, taking as a glycemia value the average of 2 measurements with an interval of 24 hours between each record
Capillary blood glucose at 14 days | At 14 days after the start of the intervention
  It will be recorded in mg/dl with a glucometer, taking as a glycemia value the average of 2 measurements with an interval of 24 hours between each record
Capillary blood glucose at 26 days | At 26 days after the start of the intervention
  It will be recorded in mg/dl with a glucometer, taking as a glycemia value the average of 2 measurements with an interval of 24 hours between each record

OTHER OUTCOMES:
Effectiveness of blinding | At 14 days after the start of the intervention
  The participants, evaluators and those who apply the intervention will be asked if they know the research group to which the study subject belongs.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Avendaño Coy, PhD, Study Director — University of Castilla-La Mancha
Locations (1):
- Juan Avendaño-Coy, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No